CLINICAL TRIAL: NCT02036567
Title: Longitudinal Observational Pilot Study to Assess the Capabilities of an Experimental Device to Objectively Measure Pain.
Brief Title: Evaluation of Pain Measurement Device
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alexander Zacharias Tzabazis, Principle Investigator, Stanford University
Other Study IDs: 28503
Record Dates: First submitted 2014-01-08; First posted 2014-01-15 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- surgical patients: no interventions, observational study
- laboring women: no interventions, observational study
- volunteers: pain induction by noxious heat stimulation, measurement of pain by device and documentation of pain reported by subjects

SUMMARY:
This longitudinal observational study will attempt to objectively measure pain with an experimental, non-invasive device. Patients and volunteers will receive a baseline screening with psychophysical tests and questionnaires. Investigators will apply the device to measure pain during routine clinical care and correlate patients pain ratings and analgesia requirements to that measured by the device. A more standardized approach with experimental pain stimuli will be pursued in human volunteer studies.

ELIGIBILITY:
Inclusion Criteria:

* age 18-100 years

Exclusion Criteria:

* inability to sign consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women of all ethnicities will be included.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
correlation between pain as measured by the device and reported pain and clinical events, respectively | average 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Z Tzabazis, MD, Principal Investigator — Stanford University
Locations (1):
- Department of Anesthesia, Pain and Perioperative Medicine, Stanford, California, United States